CLINICAL TRIAL: NCT03989557
Title: A Study of Platelet Function Test in the Application of Prevention of Ischemic Events After Stent Placement in Intracranial Aneurysms
Brief Title: Application of Platelet Function Test in Prevention of Ischemic Events After Stent Placement in Intracranial Aneurysms
Acronym: APISIA Trail
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNI-2019002
Record Dates: First submitted 2019-06-16; First posted 2019-06-18 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-06

CONDITIONS: Unruptured Intracranial Aneurysm; Stents; Antiplatelet Drugs
Keywords: Platelet function test; high platelet reactivity; light transmittance platelet aggregometry
MeSH Terms: interventions — Aspirin; Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monitoring Arm (Experimental): Randomization: based on light transmittance aggregometry, modified dose of antiplatelet therapy(aspirin and ticagrelor) was used for high platelet reactivity(HPR) patients with intracranial stent placement, and standard antiplatelet regimen(aspirin and clopidogrel) was used in non-HPR patients.
  Interventions: Drug: Aspirin and clopidogrel/Ticagrelor; Device: Light transmittance aggregometry
- Conventional Arm (Experimental): Randomization: without light transmittance aggregometry, standard antiplatelet regimen was used for unruptured aneurysm patients with intracranial stent.
  Interventions: Drug: Aspirin and clopidogrel/Ticagrelor

INTERVENTIONS:
Drug: Aspirin and clopidogrel/Ticagrelor — The modification of aspirin and clopidogrel/ticagrelor maintenance doses based on a biomarker assays.
  Arms: Monitoring Arm
Device: Light transmittance aggregometry — point-of-care method to assess platelet function by light transmittance aggregometry.
  Arms: Monitoring Arm
Drug: Aspirin and clopidogrel/Ticagrelor — maintenance dose of aspirin, clopidogrel and ticagrelor.

SUMMARY:
This study was designed to identify high platelet reactivity (HPR) who might have in-stent thrombosis in unruptured aneurysm with intracranial stent placement with light transmittance platelet aggregometry (LTA). For HPR patients, higher ischemic stroke rate maybe occurred, and we hypothesis that dose adjustment of aspirin and clopidogrel based on LTA monitoring maybe reduces the rate of ischemic stroke compared to a standard strategy after intracranial stent implantation at early periprocedural period and 1 month follow-up period.

DETAILED DESCRIPTION:
For the patients of unruptured intracranial aneurysms with stent placement, standard antiplatelet therapy (100mg aspirin + 75mg clopidogrel) is considered to be the most effective antiplatelet regimen in reducing ischemic complications. However, despite the use of standard antiplatelet therapy, a number of patients continue to have ischemic events. A hypothesis is that high platelet reactivity (HPR) patients identified by platelet function test have higher ratio of the ischemic events, and dose adjustment of HPR patients reduces the rate of the ischemic complications at early periprocedural period and follow-up period.

Objectives: The study aim to evaluated the superiority of the strategy of platelet function test(Monitoring Arm) with the modified strategy in HPR patients compared to the standard strategy (Conventional Arm) whether reduce the primary endpoint after intracranial stent implantation at early periprocedural period (7 days) and 1 months follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80, male or non-pregnant female;
2. patients have unruptured aneurysm who plan to undergo intracranial stent placement;
3. patients with less than 2 of modified Rankin scale score at the day of enrollment;
4. patients who is able to understand the objective of the trial, agrees and signs the written informed consent form.

Exclusion Criteria:

1. The complications related to operation or material quality, such as guidewire pierces out blood vessel, coil herniation, incompletely opened stent, etc;
2. Simultaneous treatment of other cerebrovascular diseases, such as intracranial arteriovenous malformation, Intracranial arteriovenous fistula, etc;
3. Patient with history of hypersensitivity of aspirin, clopidogrel, or ticagrelor;
4. Patients with preoperative prophylactic use of tirofiban;
5. Patients with a high possibility of active bleeding, such as symptomatic intracranial hemorrhage or active gastric ulcer; or patients with coagulopathy;
6. Patients with thrombocytopenia (platelet count <100,000/mm3 within three months before enrollment);
7. patient using anticoagulant;
8. Pregnant or lactating women;
9. Patients with malignant diseases, such as liver disease, kidney disease, congestive heart failure, malignant tumors, etc;
10. Poor compliance patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-08-13 (Actual)

PRIMARY OUTCOMES:
A thromboembolic event during the early periprocedural period (within 7 days after stent placement) | within 7 days of patients' enrolled.
  The thromboembolic events were assessed by clinical examination. The thromboembolic events was a composite of ischemic stroke, transient ischemic attack, stent thrombosis, urgent revascularization, myocardial infarction, cerebrovascular death.

SECONDARY OUTCOMES:
A thromboembolic event during the 1 month follow-up periods. | within 1 month of patients' enrolled.

OTHER OUTCOMES:
Major bleeding and minor bleeding | within 1 month of patients' enrolled.
  Bleeding complications were accorded to Thrombolysis in Myocardial Infarction (TIMI) bleeding criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Neurosurgical Institute and Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li W, Zhu W, Wang A, Zhang G, Zhang Y, Wang K, Zhang Y, Wang C, Zhang L, Zhao H, Wang P, Chen K, Liu J, Yang X. Effect of Adjusted Antiplatelet Therapy on Preventing Ischemic Events After Stenting for Intracranial Aneurysms. Stroke. 2021 Dec;52(12):3815-3825. doi: 10.1161/STROKEAHA.120.032989. Epub 2021 Sep 20. PMID 34538087